CLINICAL TRIAL: NCT03863106
Title: The Lyon Real World Evidence in Metastatic NeuroEndocrine Tumours
Acronym: LyREMeNet
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: LyREMeNet
Record Dates: First submitted 2018-09-27; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Gastro-enteropancreatic Neuroendocrine Tumor; Health Care Costs; Metastatic Cancer
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Metastatic gastroenteropancreatic and lung neuroendocrine tumors — Patients with metastatic GEP and lung NETs will be selected via the Cancer Database on NEN of the Hospices Civils de Lyon. Data from this database will be matched with the French nationwide claims and hospitalization database (SNDS database), allowing access to the corresponding healthcare resources use and their related costs. Data regarding clinical and tumour characteristics and treatments patterns will be collected via the database between 1 January 1990 and 31 of December 2017.
  Other Names: Metastatic NETs population description Healthcare resources use and related cost Clinical parameter: Demographic and tumour characteristics, treatments patterns

SUMMARY:
Neuroendocrine tumours (NETs) are rare and include a heterogeneous group of neoplasms derived from the endocrine system found in the gastrointestinal tract, pancreas and lung. Gastroenteropancreatic (GEP) NETs represent the majority of neuroendocrine neoplasms (NEN) and the annual incidence of all GEP-NETs has been estimated to 6.98 per 100,000 person-years in 2012 and is steadily rising. While data on the incidence of metastatic GEP-NET is limited, more than 50% of patients with GEP-NET have metastatic disease at the time of diagnosis. Incorrect and delayed diagnoses are still common. Treatment options include surgery, locoregional interventions, and systemic treatment.

The Lyon Real world Evidence in Metastatic NeuroEndocrine Tumours study (LyREMeNET) is a descriptive observational cohort study. The main objective is to assess the healthcare resources use and the corresponding costs for management of patients with metastatic GEP and lung NETs. The secondary objective is to describe the clinical characteristics, prognostic factors, treatment patterns, and the overall survival among patients with metastatic GEP and lung NETs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of well-differentiated metastatic neuroendocrine tumour (either synchronous or metachronous)
* Diagnosis performed between 1 January 1990 and 31 December of 2017
* Patients seen at least once at the oncologic department of Hospices Civils de Lyon.

Exclusion Criteria:

* Poorly differentiated neuroendocrine carcinoma
* Histologic mixed neuroendocrine tumour

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with i) a diagnosis of metastatic NET, either synchronous or metachronous, ii) between 1 January 1990 and 31 December of 2017, and iii) seen in the Hospices Civils de Lyon.
Sampling Method: Non-Probability Sample
Enrollment: 880 (Estimated)
Dates: Start 2017-07-15 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Cost in euros per year of healthcare resources related to the management of metastatic NETs patients. | The cost will be calculated, per year, from the date of metastatic diagnosis of NETs to the date of death or last follow-up (study end in September 2018)

SECONDARY OUTCOMES:
Treatments patterns in metastatic NETs patients | From diagnosis until first occurrence of each treatment, through study completion, estimated on september 2018
  Number of interventional and systemic treatments
Treatments patterns in metastatic NETs patients | From diagnosis until first occurrence of each treatment, through study completion, estimated on september 2018
  Cumulative duration in months of systemic treatments
Overall survival | From the date of metastatic diagnosis of NETs to the date of death or last-follow-up, through study completion, estimated on september 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Derived] Lemelin A, Maucort-Boulch D, Castel-Kremer E, Forestier J, Hervieu V, Lorcet M, Boutitie F, Theillaumas A, Robinson P, Duclos A, Lombard-Bohas C, Walter T. Elderly Patients with Metastatic Neuroendocrine Tumors Are Undertreated and Have Shorter Survival: The LyREMeNET Study. Neuroendocrinology. 2020;110(7-8):653-661. doi: 10.1159/000503901. Epub 2019 Oct 7. PMID 31586998